CLINICAL TRIAL: NCT00004890
Title: Phase IB Open-Label Rising-Dose Study of Biomed 101 in Patients Treated With Interleukin-2 for Malignancy
Brief Title: Biomed 101 and Interleukin-2 in Treating Patients With Kidney Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioMedicines (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067566; UCLA-9908051; BIOMED-101-CLP-01; NCI-G00-1708
Record Dates: First submitted 2000-03-07; First posted 2003-12-16 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2008-01

CONDITIONS: Drug Extravasation; Kidney Cancer
Keywords: stage I renal cell cancer; stage II renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer; drug extravasation
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin
Drug: Biomed 101

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill kidney cancer cells. Biomed 101 may protect normal cells from the side effects of interleukin-2.

PURPOSE: Phase I trial to study the effectiveness of Biomed 101 in treating patients receiving interleukin-2 for kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the safety and maximum tolerated dose of Biomed 101 in patients with renal cell cancer currently treated with interleukin-2 (IL-2). II. Evaluate the effect of different doses of Biomed 101 on the incidence and severity of IL-2 related toxicities and on the incidence and frequency of IL-2 dose reduction due to IL-2 induced toxicity.

OUTLINE: This is a dose escalation study of Biomed 101. Patients receive oral Biomed 101 three times daily, followed by interleukin-2 IV on days 1-5 and 16-20. Cohorts of 5 patients receive escalating doses of Biomed 101 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 5 patients experience dose limiting toxicities. Patients are followed for 1 month.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed renal cell cancer No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: At least 12 weeks Hematopoietic: WBC at least 2,000/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Hepatic: No hepatic failure No encephalopathy Bilirubin no greater than 2.5 times upper limit of normal (ULN) AST or ALT no greater than 2.5 times ULN Renal: No renal dysfunction requiring dialysis for greater than 72 hours Creatinine no greater than 2.0 mg/dL Cardiovascular: No history of sustained ventricular tachycardia (greater than 5 beats) No uncontrolled cardiac rhythm disturbances No recurrent chest pain with echocardiogram changes No angina No myocardial infarction No pericardial tamponade No moderate or severe coronary artery disease (New York Heart Association class 3 or 4) Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No significant neurological dysfunction including seizure or clinical signs of other significant neurological disease No gastrointestinal bleeding requiring surgery No concurrent infection requiring antimicrobial therapy No bowel ischemia or perforation

PRIOR CONCURRENT THERAPY: At least 30 days since prior investigational drugs No other concurrent investigational drugs No intubation required for greater than 72 hours No prior enrollment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Figlin, MD, FACP, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States